| Division | • | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | • | Reporting and Analysis Plan (RAP) |

Title: Reporting and Analysis Plan for GSK2983559 First time in human study 205021: A single-centre, randomised, double-blind (sponsor open), placebo controlled study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of GSK2983559, in single (in both fed and fasted states) and repeat oral doses in healthy participantsCompound Number: GSK2983559Effective Date: 25-NOV-2019

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 2017N322016 02.
- This RAP is intended to describe the safety, tolerability, pharmacokinetics, and pharmacodynamics of GSK2983559, in single (in both fed and fasted states) and repeat oral doses in healthy participants.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverables.

### **RAP Author(s):**

| Approver | Date | Approval Method |
|---|---|---|
| Statistics Leader (II Biostatistics) | 14-Oct-2019 | Author/Email |
| Programming Manager (II Clinical Programming) | 17-Oct-2019 | Email |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Scientist Director (II Discovery Medicine) | 14-Oct-2019 | Email |
| Director (II Clinical Pharmacology Modelling & Simulation) | 17-Oct-2019 | Email |
| Global Clinical Development Manager (II Global Clinical Sciences and Delivery) | 15-Oct-2019 | Email |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Senior Statistics Director (II Clinical Statistics) | 25-Nov-2019 | eSignature CARS |
| Programming Manager (II Clinical Programming) | 22-Nov-2019 | eSignature CARS |

# **TABLE OF CONTENTS**

| | | P | AGE |
|---|---|---|---|
| 1. | INTROD | UCTION | 5 |
| 2. | 2.1. C<br>2.2. St<br>2.3. St | RY OF KEY PROTOCOL INFORMATION thanges to the Protocol Defined Statistical Analysis Plan tudy Objective(s) and Endpoint(s). tudy Design tatistical Hypotheses / Statistical Analyses | 5<br>6 |
| 3. | 3.1. In | D ANALYSESterim Analysesinal Analyses | 11 |
| 4. | | IS POPULATIONSrotocol Deviations | |
| 5. | CONVEN | ERATIONS FOR DATA ANALYSES AND DATA HANDLING NTIONStudy Treatment & Sub-group Display Descriptors | 13 |
| | 5.2. Ba | aseline Definitions | 13<br>14 |
| | 5.5. M<br>5.6. O | Iultiple Comparisons and Multiplicity Sther Considerations for Data Analyses and Data Handling Conventions | 14 |
| 6. | | POPULATION ANALYSES Overview of Planned Study Population Analyses | |
| 7. | 7.1. A | ANALYSESdverse Events Analyseslinical Laboratory Analysesbther Safety Analyses | 17<br>17 |
| 8. | 8.1. P | ACOKINETIC ANALYSESrimary Pharmacokinetic Analyses | 18<br>18<br>18 |
| | 8.<br>8.<br>8.2. Se | 1.2. Summary Measures | 19<br>19<br>19<br>20 |
| | 8. | .2.2. Summary Measure | 20 |
| a | | ACODYNAMIC ANALYSES | 21 |

### CONFIDENTIAL

| 2 | 0.5 | · ^ · | 2 |
|---|-----|-------|---|
| | US | NJ. | / |

| | 9.1. | | ory Pharmacodynamic Analyses | |
|---|---|---|---|---|
| | | 9.1.1. | Endpoint / Variables | |
| | | 9.1.2. | Summary Measure | |
| | | 9.1.3. | Population of Interest | 2 1 |
| 10. | REFE | RENCES. | | 22 |
| 11. | | | | 23 |
| | 11.1. | Appendix | x 1: Protocol Deviation Management and Definitions for Per | |
| | 44.0 | Protocol | Population | 23 |
| | 11.2. | Appendix | x 2: Schedule of Activities | 24 |
| | 11.0 | | Protocol Defined Schedule of Events | |
| | 11.3. | 11.3.1. | x 3: Assessment Windows Definitions of Assessment Windows for Analyses | |
| | 11.4. | _ | x 4: Study Phases and Treatment Emergent Adverse | 20 |
| | 11.4. | | | 27 |
| | | 11.4.1. | Study Phases | |
| | | 11.7.1. | 11.4.1.1. Study Phases for Concomitant Medication | |
| | | 11.4.2. | Treatment Emergent Flag for Adverse Events | |
| | 11.5. | | x 5: Data Display Standards & Handling Conventions | |
| | | 11.5.1. | Reporting Process | 29 |
| | | 11.5.2. | Reporting Standards | |
| | | 11.5.3. | Reporting Standards for Pharmacokinetic | |
| | 11.6. | Appendix | x 6: Derived and Transformed Data | |
| | | 11.6.1. | General | |
| | | 11.6.2. | Study Population | |
| | | 11.6.3. | Safety | |
| | 11.7. | | x 7: Reporting Standards for Missing Data | |
| | | 11.7.1. | | |
| | | 11.7.2. | Handling of Missing Data | |
| | 11.8. | Annondi | 11.7.2.1. Handling of Missing and Partial Datesx 8: Values of Potential Clinical Importance | |
| | 11.0. | 11.8.1. | Laboratory Values | |
| | | 11.8.2. | ECG | |
| | | 11.8.3. | | |
| | 11.9. | | x 9: Abbreviations & Trade Marks | |
| | | | Abbreviations | |
| | | 11.9.2. | | |
| | 11.10. | Appendix | x 10: List of Data Displays | |
| | | | Data Display Numbering | |
| | | | Mock Example Shell Referencing | |
| | | | Deliverables | |
| | | | Study Population Tables | |
| | | | Safety Tables | |
| | | | Safety Figures | |
| | | | Pharmacokinetic Tables | |
| | | | Pharmacokinetic Figures | |
| | | | PharmacodynamicTables | |
| | | | .Pharmacodynamic Figures | |
| | | | .ICH Listings | |
| | | 11.10.12 | . 1 NOTE TO LESTINGS | 00 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 205021:

| Revision Chronology: | | |
|---|---|---|
| 2017N322016_00 | 06-OCT-2017 | Original |
| 2017N322016_01 | 17-OCT-2017 | Original Protocol Republishing |
| 2017N322016_02 | 24-JUL-2018 | Formulation change to enteric capsule |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

This study was terminated during Cohort 2 of Part A. Participants in Cohort 2 received only 2 of 4 planned single doses.

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Part A (single dose): Dose proportionality will be assessed by visual inspection of dose normalised AUC(0 ∞) [or if not available AUC(0-t)] and Cmax values versus dose. Analysis of these logetransformed parameters may be carried out, using the power model. | Summary of dose normalised PK parameters will be replaced by summary of PK parameters No analyses of log-transformed data will be conducted | Study terminated prior to<br>full dose escalation<br>completion |
| Part A (food effect): The ratio of fed state to fasted state may be assessed for the loge-transformed parameters AUC(0-∞) [or if not available AUC(0-t)] and Cmax. The effect of food will be assessed utilising a mixed effects model, with fed state (fasted or fed) as a fixed effect and participant as a random effect | No food effect summaries<br>or statistical analyses | Study terminated prior to fed dosing period |
| Part B: The extent of accumulation after repeat | No Part B summaries or<br>statistical analyses | Study terminated prior to<br>Part B multiple ascending |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| dosing, the observed accumulation ratio (Ro), may be determined. The plasma steady state ratio (Rs) and an assessment of plasma steady state across the trough concentrations may also be made. Dose proportionality may be assessed using similar methods to the single dose Part A. | | dose cohorts |
| For combined 5-ABT and NAc-5-ABT (corrected to 5-ABT), observed Cmax and Tmax will be determined using non-compartmental methods and will be summarised descriptively | 5-ABT and NAc-5-ABT (corrected to 5-ABT) concentrations will be listed. No PK parameters will be produced | Limited number of subjects<br>with quantifiable 5-ABT and<br>NAc-5-ABT PK<br>concentrations to warrant<br>summaries or PK<br>parameter derivations |
| To investigate the metabolic profile of GSK2983559 following single and/or repeat doses in healthy participants in urine | No urine data will be reported | Data is no longer planned<br>due to study termination<br>prior to urine samples being<br>analysed |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the safety and tolerability of single (fed and fasted) and repeat doses of GSK2983559 in healthy participants. Secondary Objectives | <ul> <li>Safety and tolerability of GSK2983559 as<br/>assessed by clinical monitoring and reporting of<br/>adverse events and serious adverse events,<br/>change in laboratory values, ECG, vital signs,<br/>physical examinations.</li> <li>Secondary Endpoints</li> </ul> |
| To characterise the PK profile of single (fasted) doses of GSK2983559 and its active moiety GSK2668176 in healthy participants. | Derived PK parameters for GSK2983559 and GSK2668176 including area under the plasma drug concentration versus time curve (AUC <sub>(0-t)</sub> , AUC <sub>(0-∞)</sub> ), maximum observed plasma drug concentration (C <sub>max</sub> ), time to maximum observed plasma drug concentration (t <sub>max</sub> ), and terminal half-life (t <sub>1/2</sub> ) following single (fasted) doses, where data allow. |
| To characterise the PK profile of repeat doses of GSK2983559 and its active | <ul> <li>Derived PK parameters for GSK2983559 and<br/>GSK2668176 including area under the plasma<br/>drug concentration versus time curve (AUC<sub>(0-t)</sub>,</li> </ul> |

| Objectives | Endpoints |
|---|---|
| moiety GSK2668176 in healthy participants. | AUC <sub>(0-т)</sub> ), maximum observed plasma drug concentration (C <sub>max</sub> ), time to maximum observed plasma drug concentration (t <sub>max</sub> ), and terminal half-life (t <sub>1/2</sub> ) following single and repeat doses, and estimation of an accumulation ratio where data allow. |
| To assess the effect of food on<br>the pharmacokinetics of<br>GSK2983559 and its active<br>moiety GSK2668176 in fasted<br>and fed state in healthy<br>participants. | <ul> <li>Derived PK parameters for GSK2983559, and GSK2668176 including area under the plasma drug concentration versus time curve (AUC<sub>(0-t)</sub>, AUC<sub>(0-∞)</sub>), maximum observed plasma drug concentration (C<sub>max</sub>), time to maximum observed plasma drug concentration (t<sub>max</sub>), and terminal half-life (t<sub>1/2</sub>) following single (fed and fasted) dose, where data allow.</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To determine the PD effect of single and repeat doses of GSK2983559 in healthy participants. | <ul> <li>PD/biomarker endpoints may include, but not be<br/>limited to, assessments of pharmacologic effects<br/>through measurements of target engagement<br/>and pathway activation. These may include<br/>measurements of RIP-2 receptor occupancy,<br/>and levels of MIP1α, MIP1β and TNF proteins,<br/>following stimulation of whole blood, as data<br/>permit. (Cohort 1 subjects only)</li> </ul> |
| To investigate the metabolic profile of GSK2983559 following single and/or repeat doses in healthy participants in blood and urine | <ul> <li>Identification and quantitative estimates of<br/>GSK2983559 and its active moiety GSK2668176<br/>and potential metabolites following single and<br/>repeat doses in plasma and urine.</li> </ul> |
| <ul> <li>To characterize exposure to 5-<br/>ABT and NAc-5-ABT after<br/>single and repeated doses of<br/>GSK2983559 in healthy<br/>participants.</li> </ul> | <ul> <li>Concentration of 5-ABT and NAc-5-ABT<br/>(adjusted to 5-ABT concentration based on<br/>molecular weight (MW)) and derive Cmax for the<br/>combined concentration curve of 5-ABT and MW<br/>adjusted NAc-5-ABT</li> </ul> |

### 2.3. Study Design



| Overview of S | Study Design and Key Features – Part A Single Ascending Dose |
|---|---|
| | 2 participants in a 7:1 and 4:1 ratios (GSK2983559: placebo) for Cohorts 1 and 2, |
| | respectively |
| Time & | Refer to Appendix 2: Schedule of Activities |
| Events | |
| Treatment<br>Assignmen<br>t | <ul> <li>At screening a unique number (case report form [CRF] number) will be assigned to<br/>any participant who has at least one Screening procedure performed, other than<br/>signed informed consent. The unique number will be used to identify individual<br/>participants during the course of the study.</li> </ul> |
| | <ul> <li>Participants who meet the screening eligibility criteria will be randomised to a treatment group through an Interactive Response Technology (IRT). The IRT will confirm the participants CRF number and provide the randomisation number, where, a randomisation number will be assigned from a randomisation schedule generated by Clinical Statistics, prior to the start of the study, using validated internal software. Once assigned, this number must not be reassigned to any other participant in the study.</li> </ul> |
| | The randomisation is centrally controlled by the IRT. |
| | Part A |
| | Within Cohort 1, participants will be assigned to one of 5 dosing sequences in a 1:1:1:1:1 ratio. |
| | Within Cohort 2, participants will be assigned to one of up to 4 dosing sequences in a 1:1:1:1 ratio. |
| | Cohort 1 Cohort 2 |
| | Sequence PBCDE PGHIJ |
| | APCDE FPHIJ |
| | ABPDE FGPIJ |
| | ABCPE FGHPJ |
| | ABCDP |
| | Participants will be randomised |
| | to: |

| Treatment code | Original Planned<br>Treatment Description | Cohort 1 Actual<br>Treatment & Cohort 2<br>Planned Treatment<br>Description |
|---|---|---|
| A | 2 mg GSK2983559 | |
| В | 10 mg GSK2983559 | 4 mg GSK2983559 |
| C | 30 mg GSK2983559 | 10 mg GSK2983559 |
| D | 75 mg GSK2983559 | 30 mg GSK2983559 |
| E | 150 mg GSK2983559 | 100 mg GSK2983599 |
| F | 300 mg GSK2983559 | 200 mg GSK2983599 |
| G | 600 mg GSK2983559 | 400 mg GSK2983559 |
| H | 800 mg GSK2983559 | 600 mg GSK2983559 |
| I | Dose TBC GSK2983559 | Dose TBC GSK2983559 |
| J | GSK2983559 Fed | GSK2983559 Fed |
| P | Placebo | |
| | were conducted due to study te | |

| Overview of S | Overview of Study Design and Key Features – Part B Multiple Ascending Dose | |
|---|---|---|
| | <ul> <li>Study terminated prior to Part B start, please refer to protocol for exact<br/>details</li> </ul> | |
| Treatment Assignment | <ul> <li>Part B treatment codes were planned to be:</li> </ul> | |
| 3 | Treatment code | Treatment Description |
| | K | Dose 1 GSK2983559 |
| | L | Dose 2 GSK2983559 |
| | M | Dose 3 GSK2983559 |
| | N | Dose 4 GSK2983559 |
| | P | Placebo |
| | · | |

# 2.4. Statistical Hypotheses / Statistical Analyses

The objectives of this study are to assess the safety and tolerability of single and repeat ascending doses of GSK2983559 in healthy volunteers. No formal hypotheses will be tested.

# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

Dose escalation meetings occurred after each period in Part A and were scheduled to occur following the completion of 14 days dosing of each cohort in Part B. The decision to proceed to the next cohort and next dose strength to be studied, was made by the Dose Escalation Committee (DEC) based on assessment of blinded safety (e.g., AEs, clinical laboratory results, vital signs and ECG), active moiety (GSK2668176) pharmacokinetic and 5-ABT concentrations obtained in all participants at the prior dose level. Individual safety data (adverse events, laboratory safety tests, ECGs and vital signs) was reviewed. This study was double blind (sponsor open), where the participant, investigator and site staff will remain blinded to the treatment allocation. Sponsor open refers only to those members of the DEC as required.

Following completion of Cohort 1: Part A and before starting Cohort 2: Part A, a GSK internal safety board (independent of DEC) reviewed the emerging PK and safety data.

A formal interim analysis was due to be performed during the study on completed cohorts in Part A of the study to aid internal decision making only. The study was terminated prior to completion of Part A.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

All participants have completed the study as defined in the protocol or the study is terminated.

All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.

All criteria for unblinding the randomisation codes have been met.

Randomisation codes have been distributed according to RandAll NG procedures.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | Screen Failure |
| | | Population Analysed. |
| Randomised | All participants who were randomly assigned to | Age ranges |
| | treatment in the study. | |
| | This population will be based on the treatment the | |
| | participant was randomised to. | |
| Safety | All randomised participants who received at least one | All other Study |
| | dose of study treatment. | Population |
| | This population will be based on the treatment the | Safety |
| | subject actually received. | |
| | Note: Participants who were not randomised but | |
| | received at least one dose of study treatment should | |
| | be listed. | |
| Pharmacokinetic | All participants in the Safety population who had at | PK |
| (PK) | least 1 non-missing PK assessment (Non-quantifiable | |
| | [NQ] values will be considered as non-missing | |
| | values). | |
| | This population will be based on the treatment the | |
| | participant actually received. | |

Refer to Appendix 10: List of Data Displays which details the population used for each display.

### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan Version 2 (08-Feb-2018).

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG | Data Display | ys for Reporting |
| Code | Description | Description | Order in TLF |
| Α | GSK2983559 single dose 1 | GSK 2 mg | 2 |
| В | GSK2983559 single dose 2 | GSK 4 mg | 3 |
| С | GSK2983559 single dose 3 | GSK 10 mg | 4 |
| D | GSK2983559 single dose 4 | GSK 30 mg | 5 |
| E | GSK2983559 single dose 5 | GSK 100 mg | 6 |
| F | GSK2983559 single dose 6 | GSK 200 mg E | 7 |
| G | GSK2983559 single dose 7 | GSK 400 mg E | 8 |
| Н | GSK2983559 single dose 8 | GSK XX mg E [1] | Not used |
| 1 | GSK2983559 single dose 9 | GSK XX mg E [1] | Not used |
| J | GSK2983559 fed single dose | Not Used | Not used |
| Р | Placebo single dose | Placebo | 1 |
| K | GSK2983559 repeat dose 1 | Not Used | Not used |
| L | GSK2983559 repeat dose 2 | Not Used | Not used |
| М | GSK2983559 repeat dose 3 | Not Used | Not used |
| N | GSK2983559 repeat dose 4 | Not Used | Not used |
| Q | Placebo repeat dose | Not Used | Not used |

<sup>1.</sup> Dose level not required as the study was terminated prior to being utilised

### 5.2. Baseline Definitions

- For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.
- For Part A, baseline definitions defined in the table are applicable to each treatment period.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing. The mean of triplicate measurements at any given time point will be used as the value for that time point unless otherwise stated.

| Parameter | Study Asses | Baseline Used in | | |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Safety | | | | |
| Clinical Chemistry/<br>Haematology/<br>Urinalysis | X | Х | X | Day 1 |
| 12-lead ECG | Х | <b>X</b> [1] | X [1] | Day 1 |
| Vital Signs | Х | Х | X [1] | Day 1 |
| Pharmacokinetic | | | • | |
| PK Concentrations | | | Х | Day 1 |
| Pharmacodynamic | | | | |
| PD Blood sample | | | Х | Day 1 |
| Target Engagement sample | | | Х | Day 1 |

<sup>[1]</sup> ECG/Vital signs recordings will be performed in triplicate at visit. Use the mean of the triplicate measurements.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

### 5.3. Multicentre Studies

This is a single centre study.

# 5.4. Examination of Covariates, Other Strata and Subgroups

There are no covariates, strata or subgroups to be investigated in this study.

# 5.5. Multiple Comparisons and Multiplicity

No adjustments for multiplicity will be required.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 11.3 | Appendix 3: Assessment Windows |
| 11.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 11.6 | Appendix 6: Derived and Transformed Data |
| 11.7 | Appendix 7: Reporting Standards for Missing Data |
| 11.8 | Appendix 8: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Screened" or "Randomised" population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

### 7. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

# 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

## 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 10: List of Data Displays.

## 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 10: List of Data Displays.

### 8. PHARMACOKINETIC ANALYSES

# 8.1. Primary Pharmacokinetic Analyses

### 8.1.1. Endpoint / Variables

PK plasma concentration-time data for the prodrug GSK2983559 and active moiety GSK2668176 will be listed, no statistical analysis will be conducted. Summary statistics of the prodrug GSK2983559 and active moiety GSK2668176 concentrations by nominal blood sampling time will be determined.

PK data will be summarised for Parts A by randomised treatment.

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 11.5.3 Reporting Standards for Pharmacokinetic).

### **Overview of Planned Pharmacokinetic Analyses**

| Endpoints | Untrans | formed | | | Log-transformed | | |
|---|---|---|---|---|---|---|---|
| | Summai | ry | Individua | al | Summar | Ŋ | Individual |
| | Т | F | F | L | Т | F | F L |
| Pharmacokinetic | | | | | | | |
| Plasma Drug concentration | Υ | <b>Y</b> [1][2] | <b>Y</b> [1] | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Summary = represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = represents FL related to any displays of individual participant observed raw data.
- 1: Linear and Semi-Log plots will be created on the same display.
- 2: Separate Mean (± SE) and Median plots will be generated.

PK plasma concentrations for 5-ABT and N-Ac-5-ABT (adjusted to 5-ABT concentration based on molecular weight (MW)) will be listed, no statistical analysis will be conducted.

### 8.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 11.5.3 Reporting Standards for Pharmacokinetic)

#### 8.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the prodrug GSK2983559 and active moiety GSK2668176 concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-inf) | Area under the concentration-time curve extrapolated to infinity will be calculated as: AUC = AUC(0-t) + C(t) / lambda_z |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Tmax | Time to reach Cmax, determined directly from the concentration-time data |
| t1/2 | Apparent terminal half-life will be calculated as: t½ = In2 / lambda_z |

#### NOTES:

Additional parameters may be included as required.

### 8.1.2. Summary Measures

- The pharmacokinetic profile following a single dose of GSK2983559
- Derived PK parameters for GSK2983559 and active moiety GSK2668176 including area under the plasma drug concentration versus time curve (AUC<sub>(0-t)</sub>, AUC<sub>(0- $\infty$ )</sub>), maximum observed plasma drug concentration (C<sub>max</sub>), time to maximum observed plasma drug concentration (t<sub>max</sub>), and terminal half-life (t<sub>1/2</sub>) following single (fasted) doses, where data allow.
- Descriptive statistics (n, arithmetic mean, standard deviation [SD] standard error [SE], 95% CI, minimum, median and maximum) will be calculated by treatment for all PK concentrations over time and for the derived PK parameters.
- In addition, for loge-transformed PK parameter variables geometric mean, 95% CI and %CV<sub>b</sub> (100 \* √ (exp(SD<sup>2</sup>) -1)) will be provided, where the SD is the standard deviation of log-transformed data.

### 8.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

# 8.1.4. Strategy for Intercurrent (Post-Randomisation) Events

- Study completion (i.e. as specified in the protocol) was defined as completing all phases of the study including the follow-up visit.
- Withdrawn participants may be replaced in the study. Replacement participants, enrolled will be dosed with the next planned treatment of the withdrawn participant, and they will not receive any treatment that the withdrawn participant has already received with the exception of the need to increase participants numbers to obtain the minimum number of evaluable participants required for interim decisions, and to obtain data in any other treatment that is required for a valid comparison. Replacement participants will receive the required treatments in the same order as planned for the original participant.

• All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.

# 8.2. Secondary Pharmacokinetic Analyses

### 8.2.1. Endpoint / Variables

5-ABT and NAc-5-ABT (adjusted to 5-ABT concentration based on molecular weight (MW)) concentrations will be listed, no statistical analysis will be conducted.

### 8.2.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 11.5.3 Reporting Standards for Pharmacokinetic)

# 8.2.2. Summary Measure

• Listings of 5-ABT and NAc-5-ABT (adjusted to 5-ABT concentration based on molecular weight (MW)) will also be provided

# 8.2.3. Population of Interest

The secondary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

### 9. PHARMACODYNAMIC ANALYSES

# 9.1. Exploratory Pharmacodynamic Analyses

### 9.1.1. Endpoint / Variables

Levels of blood MIP1 $\alpha$ , MIP1 $\beta$  and TNF proteins will be summarised and listed by randomised treatment for Cohort 1 only. No statistical analyses will be conducted.

### 9.1.2. Summary Measure

Actual values and percentage change from baseline of blood MIP1 $\alpha$ , MIP1 $\beta$  and TNF proteins will be summarised.

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 9.1.3. Population of Interest

The secondary pharmacodynamics analyses will be based on the "Safety" population, unless otherwise specified.

# 10. REFERENCES

None

# 11. APPENDICES

# 11.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - O Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.

# 11.2. Appendix 2: Schedule of Activities

# 11.2.1. Protocol Defined Schedule of Events

# Screening and Follow Up SOA

| Procedure | Screening | Follow-up Visit | Notes |
|---|---|---|---|
| | (up to 28 days prior to Day 1) | | |
| | | | Follow-up Visit to occur approximately 7 days or 5 half lives (as |
| | | | determined from Part A PK data), whichever is longer, and no greater |
| Outpatient Visit | X | Х | than 14 days after last study drug administration. |
| Informed Consent | X | | |
| Inclusion and Exclusion Criteria | X | | |
| Medical/medication/drug/alcohol history | X | | |
| Demographics | X | | |
| | | | Additional examinations may be performed, or brief examinations |
| | | | made full examinations, by the Investigator, as deemed necessary (e.g. |
| Full Physical Examination | X | | where safety or laboratory findings indicate). |
| Brief Physical Examination | | Х | |
| Drug/alc./cotinine screen | X | | Tests include alcohol breath test, urine cotinine and drug screen. |
| HIV, Hep B and Hep C screen | X | | |
| Tuberculosis Test | X | | Conducted as standard practice of the site. |
| Serum Pregnancy Test (all females) | X | | |
| FSH and estradiol (all females) | X | | |
| Hema/Chem/Urinalysis tests | X | Х | |
| Coagulation Panel | X | | |
| Lipid panel (Part B only) | X | | |
| Height and weight | X | | |
| Holter Monitoring (24-hour) | X | | |
| 12-lead ECG | Т | Х | T= Triplicate |
| | | | Vital signs to include heart rate, blood pressure, respiration rate and |
| Vital signs | Χ | Х | temperature. |
| Concomitant Medication Review | Х | Х | |
| AE and SAE Review | | Х | |

# Part A SOA

| | 1 | | | | | Stu | dy Day | (eac | h dosii | ng ses | sion) | ) | | | | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | | | | | | | Participants to be admitted to the unit the day before dosing (Day -1), |
| Procedure | Day -1 | Day 1 (time relative to dose) See Study Reference Manual for assessment time windows | | | | | | | Day 3 | and remain in house until discharge after 48-hour post-dose | | | | | | | | | |
| | | | | 3ee 3tt | uuy ker | erenc | e iviani | iai 10 | asses | sillei | it tiiii | ie wi | illuov | vs | | | | | assessments (Day 3) are completed. |
| | | Pre dose | 0 h | 15min | 30min | 1 hr | 1.5 hr | 2 hr | 2.5 hr | 3 hr | 4hr | 5hr | 6hr | 8 hr | 10 hr | 12 hr | 24 hr | 48 hr | |
| Pregnancy test (all females) | Х | | | | | | | | | | | | | | | | | | |
| | | | | | | | | | | | | | | | | | | | Additional exams./screens may be performed, or brief exams made full |
| | | | | | | | | | | | | | | | | | | | exams. by the Investigator, as deemed necessary (e.g. where safety or |
| Brief Physical Examination | Х | | | | | | | | | | | | | | | | Х | Х | laboratory findings indicate). |
| | | | | | | | | | | | | | | | | | | | Additional assessments may be performed at the discretion of the |
| Drug/alc./cotinine screen | Х | | | 1 | | | | | | | $\vdash$ | | _ | | | | | | Investigator. Tests will be conducted within site specified standards. |
| | | | | | | | | | | | | | | | | | l | l | Non-fasted samples will be collected on Day -1 and at 8 hours on Day 1. |
| Heam/Chem/Coags/Urinalysis | X | Х | | <u> </u> | | | | | | | Н | | | Χ | | | X | X | Non-fasted chemistry only will be collected at 8 hour time point. |
| Neuro. examination | X | | | | | | | Χ | | | | | | | | | _ X | X | Continuous at least Chause neet dass. Initiate at least 15 min miss to |
| Talamatin. | | < | | | | | | | | | | | > | | | | | | Continuous at least 8 hours post-dose. Initiate at least 15 min. prior to |
| Telemetry | | | | | | | | | | | | | | | | | | | dosing |
| | | | | | | | | | | | ш | | | | | | | | Vital signs to include HR, BP, respiration rate and temperature. |
| | | | | | | | | | | | ш | | | | | | | | T = Triplicate (HR and BP only) single respiration rate and temperature. |
| | | | | | | | | | | | ш | | | | | | | | Timings will be reviewed as cohorts progress and may be adjusted to |
| | | | | | | | | | | | ш | | | | | | | | ensure appropriate measurements relative to peak concentrations for |
| Vital signs | Х | т | | | Х | | Х | х | Х | | l x l | | | х | | Х | x | х | subsequent cohorts. |
| 12-lead ECG | Т | Т | | | | | Х | Х | Х | | х | | | Х | | Х | Х | Х | |
| All | D | | | | | | | | | | Ι. | | | | | | | | Prior to dosing, participants will fast for 8 hrs overnight; no food is |
| | | | | | | | | | | | 1 | | | | | | | | allowed for at least 4 hrs post-dose. Water is permitted with dosing and |
| Meals | | | | | | | | | | | l | | F | er s | ite Sch | nedule | 2 | | at all times except 1 hour pre-dose through 2-hours post-dose. |
| | | | | | | | | | | | l | | | | | | | | Participants will receive standardized meals scheduled at the same time |
| Cohort 2, fed period | D | В | | | | | | | | | l | | | | | | | | in each period. |
| | | | | | | | | | | | | | | | | | | | A minimum interval of 30 minutes will be observed between the dosing |
| | | | | | | | | | | | | | | | | | | | of the first 2 participants at each dose level. A minimum interval of 15 |
| | | | | | | | | | | | | | | | | | | | minutes will be observed between the dosing of the remaining 6 |
| Study Treatment dosing | | | Х | | | | | | | | | | | | | | | | participants. |
| | | | | | | | | | | | | | | | | | | | The number and sampling times may be adjusted once the human PK |
| PK Blood Sample | | Х | | Х | Х | Х | Χ | Χ | Χ | Х | Х | Χ | Х | Χ | Χ | Χ | Х | Х | data are available. |
| Urine Collection for | | | | | | | | | | | | | | | | | | | Participants will void bladder prior to dosing, a sample will be kept as |
| Metabolites | | X <> | | | | | | | control. 0-24-hr urine samples will be collected. | | | | | | | | | | |
| | | | | | | | | | | | | | | | | | | | Two samples will be drawn at pre-dose. The PD sampling time points |
| | | | | | | | | | | | | | | | | | | | may be updated based on emerging PK data. PD samples will not be |
| PD Blood Sample | | X | | | | | | Х | | | | Х | | Χ | | | X | X | collected in the food efect part of the study. |
| TE Blood Sample | | Х | | | | | | Χ | | | | | | | TE samples will not be collected in the food effect part of the study | | | | |
| Adverse Event Review | | < | | | | | | | | -X | | | | | | | | > | See section 10.1.1 for pre-dose SAE requirements |
| Concomitant Med. | | | | | | | | X | | | | | | | | | | > | |
| For ECG and vital signs T=Triplicate, For Meals B=Breakfast, D=Dinner | | | | | | | | | | | | | | | | | | | |

# 11.3. Appendix 3: Assessment Windows

# 11.3.1. Definitions of Assessment Windows for Analyses

No Assessment Windows will be defined for Analysis, and summaries and analyses will be based on nominal visits.

# 11.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

### 11.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the start and/or stop date/time of the study treatment within the period for Part A.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date > Study Treatment Stop Date + 1 |

### 11.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 11.4.2. Treatment Emergent Flag for Adverse Events

| Flag D | Definition |
|---|---|
| Treatment • Emergent | <ul> <li>If AE onset date is on or after treatment start date &amp; on or before treatment stop<br/>date +1.</li> </ul> |
| • | For studies with greater than one treatment period (e.g., crossover study), if AE onset is during one period and worsens during a later period it would be counted in both periods. For the initial period the logic would be as above. For the later period the logic would use the treatment dates associated with the later period: |

### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 11.5. Appendix 5: Data Display Standards & Handling Conventions

# 11.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server UK1SALX00175 | |
| HARP Compound One reporting effort will be set up for this study \ arenv \ arprod \ gsk2 mid205021 \final_01 | |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to Legacy Integrated Data Standards Library (IDSL) GSK<br/>A&amp;R dataset standards</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be | RTF files will be generated for all tables within the final_01 reporting effort. |

### 11.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings
- All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

#### **Formats**

- All data will be reported according to the actual treatment the participant received, unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

| Unscheduled Visits | Unscheduled Visits |
|---|---|
| Unscheduled visi | <ul> <li>Unscheduled visits will not be included in summary tables and/or figures.</li> </ul> |
| All unscheduled v | visits will be included in listings. |
| Descriptive Summar | Descriptive Summary Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 11.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to PKOne Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Not applicable. |
| NONMEM/PK/PD<br>File | Not applicable |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | Not applicable |
| Pharmacokinetic Para | ameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to Standards for Handling NQ Impacted PK Parameters. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to PKOne |

### 11.6. Appendix 6: Derived and Transformed Data

#### 11.6.1. General

### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 11.3.1) the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
- Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

### 11.6.2. Study Population

### **Treatment Compliance**

Treatment compliance will be calculated based on the formula:

Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \* Frequency)

Planned Treatment Duration is defined as 1 day in Part A in each period

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Participants who were randomised but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

Cumulative Dose = Sum of (Number of Days x Total Daily Dose)

If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

### 11.6.3. Safety

### **ECG Parameters**

### **RR Interval**

- IF RR interval (msec) is not provided directly, then RR can be derived as:
  - o If QTcF is machine read, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^{3} \right] * 1000$$

If ECGs are manually read, the RR value preceding the measurement QT interval should be a

### **ECG Parameters**

collected value THEN do not derive.

### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcF will be derived as:

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1</li>

# 11.7. Appendix 7: Reporting Standards for Missing Data

# 11.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as all phases of the study including the last scheduled procedure shown in the SoA (see Appendix 2).</li> <li>Withdrawn subjects may have been replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> <li>Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits.</li> </ul> |
| Liver<br>Chemistry<br>Stopping<br>Criteria | <ul> <li>Discontinuation of study treatment for abnormal liver tests is required when: <ul> <li>in the presence of abnormal liver chemistries not meeting protocol-specified stopping rules, the investigator believes study treatment discontinuation is in the best interest of the participant.</li> <li>ALT ≥ 3 x ULN.</li> </ul> </li> <li>Note: Refer to Appendix 7 of the protocol for details of the required assessments if a participant meets the above criteria.</li> </ul> |
| QTc<br>Stopping<br>Criteria | A participant that meets either bulleted criterion based on the average of triplicate ECG readings will be withdrawn from study treatment: |
| Nervous<br>System<br>Stopping<br>Criteria | <ul> <li>A participant will be withdrawn from the study if: <ul> <li>A Grade 3 or greater CTCAE Nervous System finding is observed or a significant neurologic change from a participant's baseline physical examination is observed.</li> <li>Any adverse event included in the CTCAE for Nervous System, which is also considered to be clinically significant by the Principal Investigator, will be reviewed for potential participant withdrawal.</li> </ul> </li> </ul> |

# 11.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 11.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |

| Element | Reporting Detail |
|---|---|
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 11.8. Appendix 8: Values of Potential Clinical Importance

# 11.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | D. ". ( | Male | | 0.54 |
| Hematocrit | Ratio of | Female | | 0.54 |
| | ' | $\Delta$ from BL | ↓0.075 | |
| | /1 | Male | | 180 |
| Haemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category Clinical Concern Range | | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Phosphorus | mmol/L | | <0.8 | >1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

# 11.8.2. ECG

| ECG Parameter | Units | Category | Clinical Concern Range | |
|---|---|---|---|---|
| | | | Lower | Upper |
| Absolute | | | | |
| Absolute QTc Interval | msec | H1 | > 450 | < 480 |
| | | H2 | ≥ 480 | ≤ 500 |
| | | H3 | > 500 | |
| Absolute PR Interval | msec | L, H | < 110 | > 220 |
| Absolute QRS Interval | msec | L, H | < 75 | > 110 |
| Change from Baseline | | | | |
| Increase from Baseline QTc | msec | H1 | > 30 | ≤ 60 |
| | | H2 | > 60 | |

Note: PCIs will be determined for QTcF. If QTcF not available, PCIs will be determined for QTcB instead

# 11.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |
| Respiratory Rate | breaths/min | ≤ 8 | ≥ 20 |
| Temperature | °C | ≤ 35.5 | ≥37.8 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |
# 11.9. Appendix 9: Abbreviations & Trade Marks

#### 11.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomisation & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |

| Abbreviation | Description |
|--------------|----------------------------|
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

#### 11.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| HARP |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |
| SAS |
| WinNonlin |

#### 11.10. Appendix 10: List of Data Displays

#### 11.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|-------------|------------|
| Study Population | 1.1 to 1.11 | |
| Efficacy | | |
| Safety | 3.1 to 3.22 | 3.1 to 3.7 |
| Pharmacokinetic | 4.1 to 4.6 | 4.1 to 4.8 |
| Population Pharmacokinetic (PopPK) | | |
| Pharmacodynamic and / or Biomarker | 6.1 | 6.1 |
| Pharmacokinetic / Pharmacodynamic | | |
| Section | Listi | ngs |
| ICH Listings | 1 to | 30 |
| Other Listings | 31 to | 37 |

#### 11.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided.

| Section | Figure | Table | Listing |
|------------------------------------|----------|----------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Population Pharmacokinetic (PopPK) | POPPK_Fn | POPPK_Tn | POPPK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 11.10.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 11.10.4. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1.1. | Safety | ES8A | Summary of Subject Status and Reason for Study Withdrawal:<br>Part A | ICH E3, FDAAA, EudraCT Add footnote: Note: "Subjects" is used to refer to "Participants" in all data displays to reflect GSK display standards and CDISC SDTM/ADaM standards. | SAC |
| 1.2. | Safety | ES4 | Summary of Subject Disposition at Each Study Epoch: Part A | ICH E3 Page by cohort, include treatment column for Randomised Trt Sequence and Total Column | SAC |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure: Part A | Journal Requirements | SAC |
| Protoco | Protocol Deviation | | | | |
| 1.4. | Safety | DV1 | Summary of Important Protocol Deviations: Part A | ICH E3 | SAC |

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Popula | ation Analysed | | | · | |
| 1.5. | All Subjects | SP1 | Summary of Study Populations: Part A | IDSL Add the following footnotes: [1] Subjects are included in the Randomised population if they were randomly assigned to treatment in the study. [2] Subjects are included in the Safety population if they have been randomised and received at least one dose of study treatment. [3] Subjects are included in the Pharmacokinetic population if they are in the Safety Population and a pharmacokinetic sample was obtained and analysed. | SAC |
| 1.6. | Safety | DM1 | Summary of Demographic Characteristics: Part A | ICH E3, FDAAA, EudraCT Overall and by cohort Include treatment column for randomised treatment sequence and total column | SAC |

| Study F | Population Tabl | es | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.7. | Randomised | DM11 | Summary of Age Ranges: Part A | EudraCT Only include age ranges applicable to the study ('Adult (18-64 years)' and '>=65-84 years')) Please add footnote to say that randomised population=enrolled population. Overall and by cohort Include treatment column for randomised treatment sequence and total column | SAC |
| 1.8. | Safety | DM5 | Summary of Race and Racial Combinations: Part A | ICH E3, FDA, FDAAA, EudraCT Overall and by cohort Include treatment column for randomised treatment sequence and total column | SAC |
| Prior a | nd Concomitan | t Medications | | | • |
| 1.9. | Safety | MH4 | Summary of Current/Past Medical Conditions: Part A | ICH E3 Separate summaries for Current & Past conditions, if collected. | SAC |
| 1.10. | Safety | CM1 | Summary of Concomitant Medications: Part A | ICH E3 | SAC |
| Exposu | re and Treatment | Compliance | | | |
| 1.11. | Safety | EX5 | Summary of Exposure to Study Treatment: Part A | ICH E3 | SAC |

# 11.10.5. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | e Events (AEs) | | | | |
| 3.1. | Safety | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term: Part A | ICH E3 | SAC |
| 3.2. | Safety | AE5A | Summary of All Adverse Events by Maximum Grade / Intensity by System Organ Class and Preferred Term: Part A | ICH E3 | SAC |
| 3.3. | Safety | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity: Part A | ICH E3 | SAC |
| 3.4. | Safety | AE15 | Summary of Common (>=10%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences): Part A | FDAAA, EudraCT | SAC |
| Serious | and Other Sig | nificant Adverse l | -<br>Events | | |
| 3.5. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) : Part A | FDAAA, EudraCT | SAC |
| 3.6. | Safety | AE3 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency: Part A | IDSL | SAC |
| Laborat | ory: Chemistry | / | | | |
| 3.7. | Safety | LB1 | Summary of Chemistry Changes from Baseline: Part A | ICH E3 | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.8. | Safety | LB17 | Summary of Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline: Part A | ICH E3 | SAC |
| Labora | tory: Hematolo | ду | | | · |
| 3.9. | Safety | LB1 | Summary of Hematology Changes from Baseline: Part A | ICH E3 | SAC |
| 3.10. | Safety | LB17 | Summary of Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline: Part A | ICH E3 | SAC |
| Labora | tory: Urinalysis | 5 | | | |
| 3.11. | Safety | LB1 | Summary of Urine Concentration Changes from Baseline: Part A | ICH E3 | SAC |
| 3.12. | Safety | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline: Part A | ICH E3 | |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.13. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting: Part A | IDSL | SAC |
| 3.14. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities: Part A | IDSL | SAC |
| ECG | • | , | | , | • |
| 3.15. | Safety | EG1 | Summary of ECG Findings : Part A | IDSL | SAC |
| 3.16. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category: Part A | IDSL | SAC |
| 3.17. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit: Part A | IDSL | SAC |
| 3.18. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category: Part A | IDSL | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Si | gns | | | | |
| 3.19. | Safety | VS1 | Summary of Change from Baseline in Vital Signs: Part A | ICH E3 | SAC |
| 3.20. | Safety | VS3 /<br>VS6 /<br>VS7 | Summary of Worst Case Vital Signs Results by PCI Criteria Post-Baseline Relative to Baseline: Part A | IDSL | SAC |
| Holter | | | | | |
| 3.21. | Safety | HM1 | Summary of Holter Interpretations: Part A | | SAC |
| 3.22. | Safety | HM2 | Summary of Holter Abnormalities: Part A | | SAC |

# 11.10.6. Safety Figures

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse Events | | | | | |
| 3.1. | Safety | AE10 | Plot of Common (>=10%) Adverse Events and Relative Risk: Part A | IDSL | SAC |
| Laborat | tory | | | | |
| 3.2. | Safety | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT: Part A | IDSL | SAC |
| 3.3. | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin: Part A | IDSL | SAC |
| 3.4. | Safety | SAFE_01 | Individual Profile Plots for Liver Function Tests : Part A | Page by liver function test (ALT, AST, ALKP, BILI) Scheduled & Unscheduled Visits to be presented Panel by subject Lower reference line ULN, High Reference Line PCI as y-axis allows. Label reference line clearly on figure or in legend | SAC |
| 3.5. | Safety | SAFE_02 | Box Plot of Liver Function Tests by Period: Part A | Page by liver function test (ALT, AST, ALKP, BILI) Scheduled visits only | SAC |

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.6. | Safety | SAFE_01 | Individual Profile Plots for Renal Function Tests: Part A | Page by renal function test (Blood Urea Nitrogen, Calcium, Creatinine, Gamma GT, Potassium, Sodium, Blood Glucose – fasted, Urea) Scheduled & Unscheduled Visits to be presented Panel by subject LLN and ULN to be included as y-axis allows Label reference line clearly on figure or in legend | SAC |
| 3.7. | Safety | SAFE_02 | Box Plot of Liver Function Tests by Period: Part A | Page by renal function test (Blood Urea<br>Nitrogen, Calcium, Creatinine, Gamma<br>GT, Potassium, Sodium, Blood Glucose<br>– fasted, Urea)<br>Scheduled Visits Only | SAC |

#### 11.10.7. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharmacokinetic Concentrations | | | | | |
| 4.1. | PK | PK01 | Summary of Plasma GSK2983559 Pharmacokinetic Concentration-Time Data: Part A | Include column for 95% CI. | SAC |
| 4.2. | PK | PK01 | Summary of Plasma GSK2668176 Pharmacokinetic Concentration-Time Data: Part A | Include column for 95% CI. | SAC |
| Pharma | acokinetic Para | ımaters | | | |
| 4.3. | PK | PK03 | Summary of Derived Plasma GSK2983559 Pharmacokinetic Parameters: Part A | Include columns for parameter, period, treatment, N, n, mean, 95% CI, standard deviation [SD], standard error [SE], median, minimum and maximum. | SAC |
| 4.4. | PK | PK05 | Summary of Log-Transformed Derived Plasma GSK2983559 Pharmacokinetic Parameters: Part A | Include columns for parameter, period, treatment, N, n, geometric mean, 95% CI of geometric mean, standard deviation [SD] of logged data and %CVb. Do not summarise Tmax. | SAC |
| 4.5. | PK | PK03 | Summary of Derived Plasma GSK2668176 Pharmacokinetic Parameters: Part A | Include columns for parameter, period, treatment, N, n, mean, 95% CI, standard deviation [SD], standard error [SE], median, minimum and maximum. | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.6. | PK | PK05 | Summary of Log-Transformed Derived Plasma GSK2668176 Pharmacokinetic Parameters: Part A | Include columns for parameter, period, treatment, N, n, geometric mean, 95% CI of geometric mean, standard deviation [SD] of logged data and %CVb. Do not summarise Tmax. | SAC |

# 11.10.8. Pharmacokinetic Figures

| Pharm | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acokinetic Concer | trations | | | |
| 4.1. | PK | PK16b | Individual Plasma GSK2983559 Concentration-Time Plots (Linear and Semi-log) by Subject: Part A | | SAC |
| 4.2. | PK | PK24 | Individual Plasma GSK2983559 Concentration-Time Plots (Linear and Semi-log) by Treatment : Part A | Set Y-axis maximum value close to maximum concentration for each treatment | SAC |
| 4.3. | PK | PK19 | Mean (+ SD) Plasma GSK2983559 Concentration-Time Plots (Linear and Semi-log) by Treatment: Part A | One plot / cohort | SAC |
| 4.4. | PK | PK20 | Median (Range) Plasma GSK2983559 Concentration-Time Plots (Linear and Semi-log) by Treatment: Part A | One plot / cohort | SAC |
| 4.5. | PK | PK16b | Individual Plasma GSK2668176 Concentration-Time Plots (Linear and Semi-log) by Subject: Part A | | SAC |
| 4.6. | PK | PK24 | Individual Plasma GSK2668176 Concentration-Time Plots (Linear and Semi-log) by Treatment : Part A | | SAC |
| 4.7. | PK | PK19 | Mean (+ SD) Plasma GSK2668176 Concentration-Time Plots (Linear and Semi-log) by Treatment: Part A | One plot / cohort | SAC |
| 4.8. | PK | PK20 | Median (Range) Plasma GSK2668176 Concentration-Time Plots (Linear and Semi-log) by Treatment : Part A | One plot / cohort | |

# 11.10.9. PharmacodynamicTables

| Pharma | PharmacodynamicTables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pathwa | y Activation | | | | |
| 6.1. | Safety | PD_T1 | Summary of Actual and Percentage Change from Baseline Pathway Activation Markers by Randomised Treatment | Page by TNFα, MIP-1α, MIP-1β | SAC |

### 11.10.10. Pharmacodynamic Figures

| Pharma | Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pathwa | y Activation | | | | |
| 6.1. | Safety | | Mean(+-SE) of Actual and Percentage Change from Baseline Pathway Activation Markers by Randomised Treatment | Page by TNFα, MIP-1α, MIP-1β | SAC |

# 11.10.11. ICH Listings

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure: Part A | Journal Guidelines | SAC |
| 2. | Safety | ES3 | Listing of Reasons for Study Withdrawal Part A | ICH E3 | SAC |
| 3. | Safety | SD3 | Listing of Reasons for Study Treatment Discontinuation: Part A | ICH E3 | SAC |
| 4. | Safety | BL2 | Listing of Subjects for Whom the Treatment Blind was Broken: Part A | ICH E3 | SAC |
| 5. | Safety | TA1 | Listing of Planned and Actual Treatments: Part A | IDSL | SAC |
| Protoc | ol Deviations | | | | |
| 6. | Safety<br>: Part A | DV2A | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 7. | Safety<br>: Part A | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Popula | tions Analysed | | | | |
| 8. | All Subjects<br>(Part A) | SP3a | Listing of Subjects Excluded from Any Population | ICH E3 | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 9. | Safety<br>: Part A | DM4 | Listing of Demographic Characteristics: Part A | ICH E3 Include Weight & BMI from vitals | SAC |
| 10. | Safety<br>: Part A | DM10 | Listing of Race: Part A | ICH E3 | SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | Prior and Concomitant Medications | | | | |
| 11. | Safety<br>: Part A | CP_CM4 | Listing of Concomitant Medications | IDSL | SAC |
| Exposi | re and Treatme | ent Compliance | | | |
| 12. | Safety<br>: Part A | EX4 | Listing of Exposure Data | ICH E3 | SAC |
| Advers | e Events | | | | |
| 13. | Safety<br>(Part A) | AE9CP | Listing of All Adverse Events: Part A | ICH E3 | SAC |
| 14. | Safety<br>: Part A | AE7 | Listing of Subject Numbers for Individual Adverse Events: Part A | ICH E3 | SAC |
| 15. | Safety<br>: Part A | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text: Part A | IDSL | SAC |
| Serious | s and Other Sig | nificant Adverse l | Events | | |
| 16. | Safety<br>: Part A | AE9CPa | Listing of Serious Adverse Events: Part A | ICH E3 | SAC |
| 17. | Safety<br>(Part A) | AE14 | Listing of Reasons for Considering as a Serious Adverse Event: Part A | ICH E3 | SAC |
| 18. | Safety<br>(Part A) | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment: Part A | ICH E3 | SAC |
| All Lab | oratory | | | | |
| 19. | Safety<br>: Part A | LB6 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance: Part A | ICH E3 | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 20. | Safety<br>(Part A) | LB6 | Listing of Laboratory Values of Potential Clinical Importance: Part A | | SAC |
| 21. | Safety<br>: Part A | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |
| 22. | Safety<br>: Part A | UR2B | Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| ECG | | | | | |
| 23. | Safety<br>: Part A | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | IDSL | SAC |
| 24. | Safety<br>: Part A | EG4 | Listing of ECG Values of Potential Clinical Importance | IDSL | SAC |
| 25. | Safety<br>: Part A | EG4 | Listing of All ECG Changes for Subjects with Any Value of Potential Clinical Importance | IDSL | SAC |
| 26. | Safety<br>: Part A | EG4 | Listing of ECG Changes of Potential Clinical Importance | IDSL | SAC |
| 27. | Safety<br>(Part A) | EG6 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding | IDSL | SAC |
| 28. | Safety<br>: Part A | EG6 | Listing of Abnormal ECG Findings | IDSL | SAC |
| Vital Si | gns | | | | |
| 29. | Safety<br>(Part A) | VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | IDSL | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 30. | Safety<br>(Part A) | VS5 | Listing of Vital Signs of Potential Clinical Importance | IDSL | SAC |

### 11.10.12. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharmacokinetic | | | | | |
| 31. | Pharmacokinetic | PK08 | Listing of Plasma GSK2983559 Pharmacokinetic Concentration-Time Data: Part A | | SAC |
| 32. | Pharmacokinetic | PK08 | Listing of Plasma GSK2668176 Pharmacokinetic Concentration-Time Data: Part A | | SAC |
| 33. | Pharmacokinetic | PK08 | Listing of Plasma 5-ABT Pharmacokinetic Concentration-Time Data: Part A | | SAC |
| 34. | Pharmacokinetic | PK08 | Listing of Plasma NAc-5-ABT Pharmacokinetic Concentration-<br>Time Data: Part A | | SAC |
| Pharmacodynamic | | | | | |
| 35. | Safety | | Listing of Pathway Activation Markers | TNF $\alpha$ , MIP-1 $\alpha$ , MIP-1 $\beta$ | SAC |